CLINICAL TRIAL: NCT02317562
Title: International, Multicentre, Efficacy and Safety Study of I10E in the Maintenance Treatment of Patients With Chronic Inflammatory Demyelinating Polyradiculoneuropathy: Extension of PRISM Study I10E-1302"
Brief Title: Efficacy and Safety Study of I10E in the Maintenance Treatment of Patients With CIDP: Extension of PRISM Study I10E-1302
Acronym: PRISM2
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor's decision
Sponsor: Laboratoire français de Fractionnement et de Biotechnologies (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I10E-1306
Record Dates: First submitted 2014-12-11; First posted 2014-12-16 (Estimated); Results first posted 2021-04-20 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Chronic Inflammatory Demyelinating Polyradiculoneuropathy
Keywords: Peripheral neuropathy; Disimmune disease; Neurology chronic disease; Rare disease
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating; Peripheral Nervous System Diseases; Rare Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- I10E Arm (Experimental)
  Interventions: Drug: I10E

INTERVENTIONS:
Drug: I10E — Patients who met all eligibility criteria will receive 0.5 g/kg of IMP every 3 weeks during 45 weeks.

SUMMARY:
Primary objective:

To assess the efficacy of I10E administered at a reduced maintenance dose in sustaining CIDP response after an initial 6-month treatment in PRISM study. (I10E-1302).

Secondary objective:

To assess the safety of I10E in this patient population.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patient aged 18 years or more.
2. Responder patient who have completed the last visit of PRISM I10E-1302 study defined as a patient with a decrease ≥1 point in the adjusted INCAT disability score between baseline and the end-of-study (EOS) visit of PRISM I10E-1302 study.
3. Covered by national healthcare insurance system as required by local regulations.
4. Written informed consent obtained prior to any study-related procedures.

Exclusion Criteria:

1. History of severe allergic reaction or serious adverse reaction to any Ig.
2. Known hypersensitivity to human Ig or to any of the excipients of I10E (glycine and polysorbate 80).
3. History of cardiac insufficiency (New York Heart Association (NYHA) III/IV), uncontrolled cardiac arrhythmia, unstable ischemic heart disease, or uncontrolled hypertension.
4. History of venous thromboembolic disease, myocardial infarction or cerebrovascular accident.
5. Risk factor for blood hyperviscosity such as cryoglobulinemia or haematological malignancy with monoclonal gammopathy.
6. Body mass index (BMI) ≥40 kg/m².
7. Glomerular filtration rate <80 mL/min/1.73m² measured according to the Modified Diet Renal Disease (MDRD) calculation.
8. Any other ongoing disease that may cause chronic peripheral neuropathy, such as toxin exposure, dietary deficiency, uncontrolled diabetes, hyperthyroidism, cancer, systemic lupus erythematosus or other connective tissue diseases, infection with HIV, Hepatitis B Virus (HBV) or Hepatitis C Virus (HCV), Lyme disease, multiple myeloma, Waldenström's macroglobulinaemia, amyloidosis, and hereditary neuropathy.
9. Woman with positive results on a urine pregnancy test or breastfeeding woman or woman of childbearing potential without an effective contraception.
10. Any other serious medical condition that would interfere with the clinical assessment of CIDP or use of I10E or prevent the patient from complying with the protocol requirements.
11. Increasing dosage or introduction of a systemic corticosteroids therapy within the last 3 months prior to screening, at a dose higher than 10 mg daily prednisolone or equivalent. Topical corticosteroids are permitted.
12. Treatment within 12 months prior to screening with immunomodulatory or immunosuppressant agents (including but not limited to cyclophosphamide, cyclosporine, interferon-α, interferon-β1a, anti-CD20, alemtuzumab, aziathioprine, etanercept, mycophenolate mofetil and methotrexate) or haemopoetic stem cell transplantation.
13. Plasma exchange, blood products or derivatives administered within the last 3 months prior to screening.
14. Anticipated poor compliance of patient with study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2015-11; Primary Completion 2017-07-28 (Actual); Study Completion 2017-07-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo NOBILE-ORAZIO, MD, Principal Investigator — IRCCS Instituto Clinico Humanitas, Milano, Italy
Locations (30):
- France (6):
  - CHU de Bordeaux - Hôpital Pellegrin, Bordeaux
  - Hôpital général du CHU de Dijon, Dijon
  - CHU de Nice - Hôpital l'Archet, Nice
  - CHU paris - Hôpital Pitié salpétrière, Paris
  - CHU de Saint Etienne - Hôpital Nord, Saint-Etienne
  - Hôpital de Hautepierre, Strasbourg
- Italy (7):
  - IRRCS Azienda Ospedaliera Universitaria, Genova
  - IRCCS Instituto Clinico Humanitas, Milan
  - IRRCS Istutito Nazionale Neurologico Besta, Milan
  - Ospedale San Raffaele IRCCS, Milan
  - Azienda Ospedaliera Universitaria di Padova, Padua
  - Università Cattolica del sacro Cuore, Roma
  - Azienda Ospedaliera Universitaria san Giovanni, Torino
- Spain (5):
  - Hospital de la santa creu i Sant Pau, Barcelona
  - Hospital General Universitario Gregorio, Madrid
  - Hospital Clinico Universitario de Santiago, Santiago de Compostela
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitario i Politècnico La Fe, Valencia
- Tunisia (5):
  - Tunisia Hôpital Razi, Manouba
  - Hôpital Fattouma Bourguiba, Monastir
  - Hôpital Habib Bourguiba, Sfax
  - Hôpital Sahloul, Sousse
  - Hôpital Militaire de Tunis, Tunis
- Turkey (Türkiye) (5):
  - Ankara university medical school Neurology, Ankara
  - Hacettepe University medical School Neurology, Ankara
  - Uludag University Medical School Neurology, Bursa
  - istanbul University Cerrahpasa Medical School Neurology, Istanbul
  - Marmara Universitesi Egitim Ve Arastirma Hastanesi, Istanbul
- United Kingdom (2):
  - Southhampton general Hospital, Southhampton
  - University Hospital of North Straffordshire, Straffordshire

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between 09 November 2015 and 23 June 2017, 20 subjects from 14 sites signed an informed consent.
Pre-assignment Details: 20 subjects signed an informed consent but only 19 subjects enrolled (1 screening failure).
Groups:
- I10E Arm: Participation in the study was proposed to all subjects who completed and responded to treatment in PRISM study, satisfying in eligibility criteria and were willing to continue I10E at a reduced maintenance dose.
  Each subject was expected to receive 16 doses of I10E (study drug) at 0.5 g/kg over 1 to 2 days, every 3 weeks.
Period: Overall Study
Arm/Group | I10E Arm
Started | 19
Completed | 5
Not Completed | 14
Not completed — Physician Decision | 1
Not completed — early termination of the study | 8
Not completed — Lack of Efficacy | 4
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | I10E Arm
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 4
Age, Continuous [Median (Full Range); unit: years] | 50.0 [24 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 11
  More than one race | 0
  Unknown or Not Reported | 8
Region of Enrollment [Number; unit: participants]
  Turkey | 1
  Italy | 4
  United Kingdom | 1
  France | 2
  Tunisia | 6
  Spain | 2
  Poland | 3

OUTCOME MEASURES:

1. Primary Outcome: Efficacy Endpoint : Responder Rate at End of Study (EOS) Visit
Description: Since the study was prematurely terminated and an important number of subjects early withdrawn, the responder rate is biased and consequently not interpretable.
  Responders were defined as subjects with either:
  No change or decrease in the adjusted INCAT disability score and without any change in CIDP treatment between baseline and EOS visit. OR An increase by 1 point in the adjusted INCAT disability score without requirement of any change in CIDP treatment between baseline and EOS visit.
Time Frame: week 48 (End-of-Study)
Population: Study prematurely stopped due to sponsor decision based on the relapse rate.
Measure: Count of Participants; unit: Participants
Arm/Group | I10E Arm
Number analyzed (Participants) | 19
Participants | 15

ADVERSE EVENTS:
Time Frame: The safety was assessed by recording all AEs occurring during the study, i.e. after signature of the informed consent and until the end of the study recorded. (up to 48 weeks after inclusion).
Arm/Group | I10E Arm
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 1/19
Other Adverse Events (participants affected / at risk) | 12/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | I10E Arm (N=19)
Urinary retention (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | I10E Arm (N=19)
Hypertension (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Fatigue (General disorders) | 2 (2)
Chills (General disorders) | 1 (1)
Injection site erythema (General disorders) | 1 (1)
Injection site oedema (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Conversion disorder (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1)
Post traumatic pain (Injury, poisoning and procedural complications) | 1 (1)
Blood pressure increased (Investigations) | 2 (2)
Blood lactate dehydrogenase (Investigations) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Headache (Nervous system disorders) | 3 (5)
Migraine (Nervous system disorders) | 1 (2)
Neuralgia (Nervous system disorders) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Eczema nummular (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (3)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Conjunctivitis (Infections and infestations) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1)
Infected bite (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (2)
Nasopharyngitis (Infections and infestations) | 1 (2)
Tooth abscess (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (2)

LIMITATIONS AND CAVEATS:
This study was prematurely stopped because 4 subjects relapsed among 14 enrolled and treated subjects at the time of the early assessment of study results.

LFB BIOTECHNOLOGIES judged that it was not acceptable to continue the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-05-03): https://cdn.clinicaltrials.gov/large-docs/62/NCT02317562/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-30): https://cdn.clinicaltrials.gov/large-docs/62/NCT02317562/SAP_001.pdf